CLINICAL TRIAL: NCT03034473
Title: Translational Validation Study to Examine KFO179-1 Biomarker Scores for the Prediction and Prognosis of Advanced Primary Resectable Rectal Cancer Stages UICC II-IV, With a 5-FU-based Standard Radiochemotherapy Followed by Total Mesorectal Excision.
Brief Title: Translational Validation Study to Examine KFO179-1 Biomarker Scores for the Prediction and Prognosis of Advanced Primary Resectable Rectal Cancer Stages UICC-II-IV, With a 5-Fluorouracil-based Standard Radiochemotherapy Followed by Total Mesorectal Excision.
Acronym: TransValid-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Goettingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Torsten Liersch, Prof. Dr. med., University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TransValid-KFO179/GRCSG-A; DRKS00003659 (Registry Identifier: Deutsches Register Klinischer Studien); UTN U1111-1131-9971 (Registry Identifier: WHO Registry Network)
Record Dates: First submitted 2017-01-13; First posted 2017-01-27 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: locally advanced rectal cancer; translational research; Biomarker
MeSH Terms: interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood and tissue samples during therapy (Other): Collection of blood and tissue samples during preoperative multimodal treatment (Radiochemotherapy (RCTx) followed by total mesorectal excision (TME) and Chemotherapy (CT)) in rectal cancer.
  Interventions: Other: Translational Research and multimodal treatment

INTERVENTIONS:
Other: Translational Research and multimodal treatment — Blood/biopsy samples (tumor & mucosa) are taken pretherapeutically. Blood samples (serum & plasma) are drawn at 11 time points during RCTx (e.g. for analysis of 5-FU metabolism, genomic DNA extraction). After pathohistological workup of the TME specimen, the formalin-fixed material will be transferred to the central biobank of KFO179. Blood samples (plasma & serum) will be drawn during 5y-follow-up. Treatment (based on CAO/ARO/AIO-94- and CAO/ARO/AIO-04-phase-III trials of the GRCSG):
  Preoperative RCT: 28x1.8 Gy (total: 50.4 Gy, 5 fractions per week on d1-d38) combined with 5-FU (1000 mg/m2/d) as 120 h civ during 1st and 5th week.
  TME-surgery is performed 6 weeks after RCTx. 4 to 8 weeks after surgery, patients receive either 4 cycles 5-FU (500 mg 5-FU/m2 iv, d1-5, repeat d 29-33) or 3 cycles (6 single appl.) of FOLFOX regimen [(400 mg FA/m2, 2-h civ, d 1; 100 mg oxaliplatin/m2, 2-h civ in 500 ml Glucose 5%, d 1; 2400 mg 5-FU/m2 as 46-h civ) on d1+d15, d30+d45 and d60+d75].

SUMMARY:
The objective of the TransValid-KFO179/GRCSG-Trial-A is the validation of potential biomarkers. These are predictive (Prediction of probability of response to a certain therapy) / prognostic (predicting long-term outcome) microarray-based gene expression signatures and immunohistochemically evaluated biomarkers. The evaluation was done within the KFO179 (www.kfo179.de) - the validation is implemented in this trial.

Therefore tumor material of patients undergoing standard radiochemotherapy will be analyzed from pretreatment biopsies an residual tissue from the resection specimen after surgery. This validation and the biomaterial asservation will be incorporated into clinical routine in all participating centers as a model for the treatment of solid tumors. The obtained biomarkers with a predictive and prognostic power will be used to develop an algorithm to predict patients at high risk of local and distant cancer recurrence.

DETAILED DESCRIPTION:
The objective of the TransValid-KFO179/GRCSG-Trial-A is to validate the predictive/prognostic microarray-based gene expression signatures and single gene biomarkers (including 5-Fluorouracil (FU) metabolism, apoptosis, Kirsten Rat Sarcoma (KRAS), CpGCpG island methylation phenotype (CIMP) and TGF-beta pathway), which have been established in patients treated with standard 5-FU based RCT in the GRCSG trials (e.g. the CAO/ARO/AIO-94-, CAO/ARO/AIO-04-phase III trials). This validation will be incorporated into clinical routine in all participating centers as a model for the treatment of solid tumors. If the KFO179 biomarkers are predictive at a satisfactory level in the validation set, we will propose a prediction algorithm to stratify the patient population into a "high"-risk and "low"-risk population to develop local and distant cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 85 years, inclusive
* Histologically confirmed advanced primary rectal cancer localized up to 12 cm above the anocutaneous line (determined with a rigid rectoscope), classified as T3/T4 or N+ carcinomas or with evidence for synchronous, but resectable distant metastases (liver or lung metastases)
* No specific tumor treatment except colostomy due to tumor stenosis with ileus
* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) status ≤2
* Adequate bone marrow function (WBC >3.0x10^9/L, neutrophils >1.5x10^9/L, thrombocytes >100x10^9/L, hemoglobin ≥10 g/dl)
* Adequate liver function (bilirubin ≤2.0 mg/dl, SGOT, SGPT, AP, gamma-GT < three point five fold of upper level of normal range
* serum creatinine < 1.5 mg/dl
* Written and signed informed consent indicating the understanding of the investigational nature and the study protocol.

Exclusion Criteria:

* Pregnant or lactating women
* Men and women unwilling or unable to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment
* Prolonged drug, medication or alcohol abuse
* Previous chemotherapy (up to 2 years before diagnosis of rectal cancer)
* Previous radiotherapy to the pelvic area
* Simultaneous therapy with other anti-cancer drugs
* Participation in a clinical trial in the period 30 days prior to inclusion
* Patients (man and woman) who are not able or willing to accept treatment and follow-up care according to trial protocol
* Patients (man and woman) with uncontrolled, serious physical or mental diseases, e.g.: instable cardiac disease in spite of medical treatment, myocardial infarction during the last 3 months prior to start of trial participation

  * neurological or psychiatric dysfunction including dementia or seizure disorder
  * Disseminated infection or sepsis
  * Disseminated intravascular coagulopathy
  * Symptomatic neuropathy (NCI CTC ≥2)
* Patients with secondary malignancies except basal cell carcinoma of the skin or carcinoma in situ of the cervix, which have been successfully treated. (The inclusion of patients with other tumors that were successfully treated and no recurrence within the last 3-5 years should be discussed before registration in the trial)
* Chronic diarrhea (>grade 1 according NCI CTCAE)
* Allergic reaction to platin-derivates or study medication
* Simultaneous treatment with sorivudine and analogous
* Known Dihydropyrimidine dehydrogenase deficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-08; Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with histopathologically confirmed complete remission (pCR) (ypT0N0 R0) after preoperative RCTx related to pretherapeutically determined gene expression signature predicting tumor response to RCTx. | 1 year after surgery
  The efficacy of the pretherapeutically determined response prediction using a reliable and robust panel of biomarkers (gene expression signature) is assessed by several clinicopathological parameters after preoperative RCTx and TME-surgery that indicate response and toxicity (ypN-status, pCR, tumor regression-grading, R-status, toxicity).
  Timepoint for measuring the gene expression signature is the time of diagnosis (pretreatment biopsy); several immunohistochemical biomarkers (Thymidylatesynthase, Survivin, HER-2) will be determined in the pretreatment biopsy as well as at the time of resection in the residual tumor tissue.

SECONDARY OUTCOMES:
R0-rate of resection | 30 days after surgery based on histopathological findings and reports
  The resection status will be classified by the pathologists according to the established UICC-TNM-Classification (R0 vs R1 vs R2 resection status)
post-operative 30-day mortality | 30 days after surgery
post-operative morbidity (esp. rate of anastomotic insufficiencies) | 30 days after surgery
post-operative late complications (defecation problems, anastomotic, stenoses, loss of sphincter function) | up to 5 years after surgery
Quality of TME-surgery according to M.E.R.C.U.R.Y classification | 30 days after surgery based on surgical and histopathological findings/reports
  The quality of total mesorectal excision (TME) will be classified by the surgeons (intraoperatively according to M.E.R.C.U.R.Y criteria: good vs moderat vs poor as published in national guidelines) and independently by the pathologists (on the resected specimen according to the well established M.E.R.C.U.R.Y criteria: good vs moderate vs poor).
acute and late toxicity of the chemotherapy according to the CommonToxicity Criteria of the National Cancer Institute (CTC) (vs 4.0) | up to 5 years after therapy
Disease free survival (DSF) after 2 and 3 years (local and/or distant recurrences) | up to 3 years after surgery
Cumulative incidence of local relapses and distant metastases | up to 5 years after surgery
Overall cancer specific survival (CSS) after 3 and 5 years | up to 5 years after surgery
Quality of life (QL) according to the EORTC-Questionnaire QLQ-30 (3.0) | up to 5 years after surgery
  The EORTC-Questionnaire QLQ-30 (3.0) have to be completed at the following timepoints: before first treatment (baseline), at the end of treatment (30 days after last intervention or application) and during follow-up (12, 36 and 60 months after surgical intervention). The outcome measures at the end of treatment, 12,36,60 months after surgery will be compared to baseline. EORTC-Life Quality (LQ)-Questionnaire and Wexner Score-Questionnaire will be analysed separately.
Wexner-Score-Questionnaire | up to 5 years after surgery
  The Wexner-Score-Questionnaire have to be completed at the following timepoints: before first treatment (baseline), at the end of treatment (30 days after last intervention or application) and during follow-up (12, 36 and 60 months after surgical intervention). The outcome measures at the end of treatment, 12,36,60 months after surgery will be compared to baseline. EORTC-LQ-Questionnaire and Wexner Score-Questionnaire will be analysed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Liersch, MD, Prof., Principal Investigator — University Medical Center Goettingen; Michael Ghadimi, MD, Prof., Study Director — University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Jakob C, Aust DE, Meyer W, Baretton GB, Schwabe W, Hausler P, Becker H, Liersch T. Thymidylate synthase, thymidine phosphorylase, dihydropyrimidine dehydrogenase expression, and histological tumour regression after 5-FU-based neo-adjuvant chemoradiotherapy in rectal cancer. J Pathol. 2004 Dec;204(5):562-8. doi: 10.1002/path.1663. PMID 15538739
- [Background] Ghadimi BM, Grade M, Difilippantonio MJ, Varma S, Simon R, Montagna C, Fuzesi L, Langer C, Becker H, Liersch T, Ried T. Effectiveness of gene expression profiling for response prediction of rectal adenocarcinomas to preoperative chemoradiotherapy. J Clin Oncol. 2005 Mar 20;23(9):1826-38. doi: 10.1200/JCO.2005.00.406. PMID 15774776
- [Background] Jakob C, Liersch T, Meyer W, Baretton GB, Hausler P, Schwabe W, Becker H, Aust DE. Immunohistochemical analysis of thymidylate synthase, thymidine phosphorylase, and dihydropyrimidine dehydrogenase in rectal cancer (cUICC II/III): correlation with histopathologic tumor regression after 5-fluorouracil-based long-term neoadjuvant chemoradiotherapy. Am J Surg Pathol. 2005 Oct;29(10):1304-9. doi: 10.1097/01.pas.0000170346.55304.88. PMID 16160472
- [Background] Liersch T, Meller J, Kulle B, Behr TM, Markus P, Langer C, Ghadimi BM, Wegener WA, Kovacs J, Horak ID, Becker H, Goldenberg DM. Phase II trial of carcinoembryonic antigen radioimmunotherapy with 131I-labetuzumab after salvage resection of colorectal metastases in the liver: five-year safety and efficacy results. J Clin Oncol. 2005 Sep 20;23(27):6763-70. doi: 10.1200/JCO.2005.18.622. PMID 16170184
- [Background] Rodel C, Martus P, Papadoupolos T, Fuzesi L, Klimpfinger M, Fietkau R, Liersch T, Hohenberger W, Raab R, Sauer R, Wittekind C. Prognostic significance of tumor regression after preoperative chemoradiotherapy for rectal cancer. J Clin Oncol. 2005 Dec 1;23(34):8688-96. doi: 10.1200/JCO.2005.02.1329. Epub 2005 Oct 24. PMID 16246976
- [Background] Grade M, Ghadimi BM, Varma S, Simon R, Wangsa D, Barenboim-Stapleton L, Liersch T, Becker H, Ried T, Difilippantonio MJ. Aneuploidy-dependent massive deregulation of the cellular transcriptome and apparent divergence of the Wnt/beta-catenin signaling pathway in human rectal carcinomas. Cancer Res. 2006 Jan 1;66(1):267-82. doi: 10.1158/0008-5472.CAN-05-2533. PMID 16397240
- [Background] Grade M, Becker H, Liersch T, Ried T, Ghadimi BM. Molecular cytogenetics: genomic imbalances in colorectal cancer and their clinical impact. Cell Oncol. 2006;28(3):71-84. doi: 10.1155/2006/173815. PMID 16823176
- [Background] Jakob C, Liersch T, Meyer W, Baretton GB, Schwabe W, Hausler P, Kulle B, Becker H, Aust DE. Prognostic value of histologic tumor regression, thymidylate synthase, thymidine phosphorylase, and dihydropyrimidine dehydrogenase in rectal cancer UICC Stage II/III after neoadjuvant chemoradiotherapy. Am J Surg Pathol. 2006 Sep;30(9):1169-74. doi: 10.1097/01.pas.0000213302.13435.6e. PMID 16931962
- [Background] Liersch T, Langer C, Ghadimi BM, Kulle B, Aust DE, Baretton GB, Schwabe W, Hausler P, Becker H, Jakob C. Lymph node status and TS gene expression are prognostic markers in stage II/III rectal cancer after neoadjuvant fluorouracil-based chemoradiotherapy. J Clin Oncol. 2006 Sep 1;24(25):4062-8. doi: 10.1200/JCO.2005.04.2739. PMID 16943523
- [Background] Ghadimi BM, Grade M, Monkemeyer C, Kulle B, Gaedcke J, Gunawan B, Langer C, Liersch T, Becker H. Distinct chromosomal profiles in metastasizing and non-metastasizing colorectal carcinomas. Cell Oncol. 2006;28(5-6):273-81. doi: 10.1155/2006/529190. PMID 17167180
- [Background] Rodel C, Liersch T, Hermann RM, Arnold D, Reese T, Hipp M, Furst A, Schwella N, Bieker M, Hellmich G, Ewald H, Haier J, Lordick F, Flentje M, Sulberg H, Hohenberger W, Sauer R. Multicenter phase II trial of chemoradiation with oxaliplatin for rectal cancer. J Clin Oncol. 2007 Jan 1;25(1):110-7. doi: 10.1200/JCO.2006.08.3675. PMID 17194912
- [Background] Fietkau R, Rodel C, Hohenberger W, Raab R, Hess C, Liersch T, Becker H, Wittekind C, Hutter M, Hager E, Karstens J, Ewald H, Christen N, Jagoditsch M, Martus P, Sauer R; German Rectal Cancer Study Group. Rectal cancer delivery of radiotherapy in adequate time and with adequate dose is influenced by treatment center, treatment schedule, and gender and is prognostic parameter for local control: results of study CAO/ARO/AIO-94. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):1008-19. doi: 10.1016/j.ijrobp.2006.10.020. Epub 2006 Dec 29. PMID 17197130
- [Background] Grade M, Hormann P, Becker S, Hummon AB, Wangsa D, Varma S, Simon R, Liersch T, Becker H, Difilippantonio MJ, Ghadimi BM, Ried T. Gene expression profiling reveals a massive, aneuploidy-dependent transcriptional deregulation and distinct differences between lymph node-negative and lymph node-positive colon carcinomas. Cancer Res. 2007 Jan 1;67(1):41-56. doi: 10.1158/0008-5472.CAN-06-1514. PMID 17210682
- [Background] Liersch T, Meller J, Bittrich M, Kulle B, Becker H, Goldenberg DM. Update of carcinoembryonic antigen radioimmunotherapy with (131)I-labetuzumab after salvage resection of colorectal liver metastases: comparison of outcome to a contemporaneous control group. Ann Surg Oncol. 2007 Sep;14(9):2577-90. doi: 10.1245/s10434-006-9328-x. Epub 2007 Jun 15. PMID 17570017
- [Background] Vorwerk H, Hermann RM, Christiansen H, Liersch T, Hess CF, Weiss E. A special device (double-hole belly board) and optimal radiation technique to reduce testicular radiation exposure in radiotherapy of rectal cancer. Radiother Oncol. 2007 Sep;84(3):320-7. doi: 10.1016/j.radonc.2007.06.017. Epub 2007 Aug 13. PMID 17706310
- [Background] Rodel C, Arnold D, Hipp M, Liersch T, Dellas K, Iesalnieks I, Hermann RM, Lordick F, Hinke A, Hohenberger W, Sauer R. Phase I-II trial of cetuximab, capecitabine, oxaliplatin, and radiotherapy as preoperative treatment in rectal cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 15;70(4):1081-6. doi: 10.1016/j.ijrobp.2007.07.2356. Epub 2007 Sep 19. PMID 17881150
- [Background] Jakob C, Liersch T, Meyer W, Becker H, Baretton GB, Aust DE. Predictive value of Ki67 and p53 in locally advanced rectal cancer: correlation with thymidylate synthase and histopathological tumor regression after neoadjuvant 5-FU-based chemoradiotherapy. World J Gastroenterol. 2008 Feb 21;14(7):1060-6. doi: 10.3748/wjg.14.1060. PMID 18286688
- [Background] Stoehlmacher J, Goekkurt E, Mogck U, Aust DE, Kramer M, Baretton GB, Liersch T, Ehninger G, Jakob C. Thymidylate synthase genotypes and tumour regression in stage II/III rectal cancer patients after neoadjuvant fluorouracil-based chemoradiation. Cancer Lett. 2008 Dec 18;272(2):221-5. doi: 10.1016/j.canlet.2008.07.008. Epub 2008 Aug 21. PMID 18722050
- [Background] Kalata P, Martus P, Zettl H, Rodel C, Hohenberger W, Raab R, Becker H, Liersch T, Wittekind C, Sauer R, Fietkau R; German Rectal Cancer Study Group. Differences between clinical trial participants and patients in a population-based registry: the German Rectal Cancer Study vs. the Rostock Cancer Registry. Dis Colon Rectum. 2009 Mar;52(3):425-37. doi: 10.1007/DCR.0b013e318197d13c. PMID 19333042
- [Background] Liersch T, Rothe H, Ghadimi BM, Becker H. [Individualizing treatment for locally advanced rectal cancer]. Chirurg. 2009 Apr;80(4):281-93. doi: 10.1007/s00104-008-1617-4. German. PMID 19350305
- [Background] Liersch T, Grade M, Gaedcke J, Varma S, Difilippantonio MJ, Langer C, Hess CF, Becker H, Ried T, Ghadimi BM. Preoperative chemoradiotherapy in locally advanced rectal cancer: correlation of a gene expression-based response signature with recurrence. Cancer Genet Cytogenet. 2009 Apr 15;190(2):57-65. doi: 10.1016/j.cancergencyto.2008.11.011. PMID 19380020
- [Background] Sprenger T, Rothe H, Langer C, Becker H, Liersch T. Comment on "lymph nodes after preoperative chemoradiotherapy for rectal carcinoma: number, status, and impact on survival". Am J Surg Pathol. 2009 Jul;33(7):1107; author reply 1108. doi: 10.1097/PAS.0b013e31819ca2a4. No abstract available. PMID 19390426
- [Background] Grade M, Gaedcke J, Wangsa D, Varma S, Beckmann J, Liersch T, Hess C, Becker H, Difilippantonio MJ, Ried T, Ghadimi BM. Chromosomal copy number changes of locally advanced rectal cancers treated with preoperative chemoradiotherapy. Cancer Genet Cytogenet. 2009 Aug;193(1):19-28. doi: 10.1016/j.cancergencyto.2009.03.016. PMID 19602460
- [Background] Sprenger T, Rothe H, Homayounfar K, Beissbarth T, Ghadimi BM, Becker H, Liersch T. Preoperative chemoradiotherapy does not necessarily reduce lymph node retrieval in rectal cancer specimens--results from a prospective evaluation with extensive pathological work-up. J Gastrointest Surg. 2010 Jan;14(1):96-103. doi: 10.1007/s11605-009-1057-6. Epub 2009 Oct 15. PMID 19830503
- [Background] Folprecht G, Gruenberger T, Bechstein WO, Raab HR, Lordick F, Hartmann JT, Lang H, Frilling A, Stoehlmacher J, Weitz J, Konopke R, Stroszczynski C, Liersch T, Ockert D, Herrmann T, Goekkurt E, Parisi F, Kohne CH. Tumour response and secondary resectability of colorectal liver metastases following neoadjuvant chemotherapy with cetuximab: the CELIM randomised phase 2 trial. Lancet Oncol. 2010 Jan;11(1):38-47. doi: 10.1016/S1470-2045(09)70330-4. Epub 2009 Nov 26. PMID 19942479
- [Background] Wolff HA, Gaedcke J, Jung K, Hermann RM, Rothe H, Schirmer M, Liersch T, Herrmann MKA, Hennies S, Rave-Frank M, Hess CF, Christiansen H. High-grade acute organ toxicity during preoperative radiochemotherapy as positive predictor for complete histopathologic tumor regression in multimodal treatment of locally advanced rectal cancer. Strahlenther Onkol. 2010 Jan;186(1):30-35. doi: 10.1007/s00066-009-2037-1. Epub 2009 Dec 28. PMID 20082185
- [Background] Weiss C, Arnold D, Dellas K, Liersch T, Hipp M, Fietkau R, Sauer R, Hinke A, Rodel C. Preoperative radiotherapy of advanced rectal cancer with capecitabine and oxaliplatin with or without cetuximab: A pooled analysis of three prospective phase I-II trials. Int J Radiat Oncol Biol Phys. 2010 Oct 1;78(2):472-8. doi: 10.1016/j.ijrobp.2009.07.1718. Epub 2010 Feb 3. PMID 20133081
- [Background] Gutenberg A, Gerdes JS, Jung K, Sander B, Gunawan B, Bock HC, Liersch T, Bruck W, Rohde V, Fuzesi L. High chromosomal instability in brain metastases of colorectal carcinoma. Cancer Genet Cytogenet. 2010 Apr 1;198(1):47-51. doi: 10.1016/j.cancergencyto.2009.12.006. PMID 20303014
- [Background] Sprenger T, Rothe H, Jung K, Christiansen H, Conradi LC, Ghadimi BM, Becker H, Liersch T. Stage II/III rectal cancer with intermediate response to preoperative radiochemotherapy: do we have indications for individual risk stratification? World J Surg Oncol. 2010 Apr 13;8:27. doi: 10.1186/1477-7819-8-27. PMID 20388220
- [Background] Rodel F, Reichert S, Sprenger T, Gaipl US, Mirsch J, Liersch T, Fulda S, Rodel C. The role of survivin for radiation oncology: moving beyond apoptosis inhibition. Curr Med Chem. 2011;18(2):191-9. doi: 10.2174/092986711794088362. PMID 21110807
- [Background] Sprenger T, Rodel F, Beissbarth T, Conradi LC, Rothe H, Homayounfar K, Wolff HA, Ghadimi BM, Yildirim M, Becker H, Rodel C, Liersch T. Failure of downregulation of survivin following neoadjuvant radiochemotherapy in rectal cancer is associated with distant metastases and shortened survival. Clin Cancer Res. 2011 Mar 15;17(6):1623-31. doi: 10.1158/1078-0432.CCR-10-2592. Epub 2010 Nov 30. PMID 21118954
- [Background] Rodel C, Arnold D, Becker H, Fietkau R, Ghadimi M, Graeven U, Hess C, Hofheinz R, Hohenberger W, Post S, Raab R, Sauer R, Wenz F, Liersch T. Induction chemotherapy before chemoradiotherapy and surgery for locally advanced rectal cancer : is it time for a randomized phase III trial? Strahlenther Onkol. 2010 Dec;186(12):658-64. doi: 10.1007/s00066-010-2194-2. Epub 2010 Nov 30. PMID 21136027
- [Background] Meller J, Liersch T, Oezerden MM, Sahlmann CO, Meller B. Targeting NCA-95 and other granulocyte antigens and receptors with radiolabeled monoclonal antibodies (Mabs). Q J Nucl Med Mol Imaging. 2010 Dec;54(6):582-98. PMID 21221067
- [Background] Meller B, Rave-Franck M, Breunig C, Schirmer M, Baehre M, Nadrowitz R, Liersch T, Meller J. Novel Carcinoembryonic-Antigen-(CEA)-Specific Pretargeting System to Assess Tumor Cell Viability after Irradiation of Colorectal Cancer Cells. Strahlenther Onkol. 2011 Feb;187(2):120-6. doi: 10.1007/s00066-010-2191-5. Epub 2011 Jan 24. PMID 21271227
- [Background] Danner BC, Gerdes JS, Jung K, Sander B, Enders C, Liersch T, Seipelt R, Gutenberg A, Gunawan B, Schondube FA, Fuzesi L. Comparison of chromosomal aberrations in primary colorectal carcinomas to their pulmonary metastases. Cancer Genet. 2011 Mar;204(3):122-8. doi: 10.1016/j.cancergen.2010.12.003. PMID 21504711
- [Background] Wolff HA, Conradi LC, Schirmer M, Beissbarth T, Sprenger T, Rave-Frank M, Hennies S, Hess CF, Becker H, Christiansen H, Liersch T. Gender-specific acute organ toxicity during intensified preoperative radiochemotherapy for rectal cancer. Oncologist. 2011;16(5):621-31. doi: 10.1634/theoncologist.2010-0414. Epub 2011 May 9. PMID 21558132
- [Background] Gaedcke J, Liersch T, Hess C, Becker H, Rodel C, Ghadimi BM. [Rectal cancer: current status of multimodal therapy--when and how?]. Zentralbl Chir. 2011 Aug;136(4):334-42. doi: 10.1055/s-0031-1271581. Epub 2011 Aug 23. German. PMID 21863511
- [Background] Gehoff A, Basten O, Sprenger T, Conradi LC, Bismarck C, Bandorski D, Merkelbach-Bruse S, Schneider-Stock R, Stoehr R, Wirtz RM, Kitz J, Muller A, Hartmann A, Becker H, Ghadimi BM, Liersch T, Ruschoff J. Optimal lymph node harvest in rectal cancer (UICC stages II and III) after preoperative 5-FU-based radiochemotherapy. Acetone compression is a new and highly efficient method. Am J Surg Pathol. 2012 Feb;36(2):202-13. doi: 10.1097/PAS.0b013e31823fa35b. PMID 22251939
- [Background] Rodel C, Hofheinz R, Liersch T. Rectal cancer: state of the art in 2012. Curr Opin Oncol. 2012 Jul;24(4):441-7. doi: 10.1097/CCO.0b013e328352ea02. PMID 22450150
- [Background] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Background] Rodel C, Liersch T, Becker H, Fietkau R, Hohenberger W, Hothorn T, Graeven U, Arnold D, Lang-Welzenbach M, Raab HR, Sulberg H, Wittekind C, Potapov S, Staib L, Hess C, Weigang-Kohler K, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R; German Rectal Cancer Study Group. Preoperative chemoradiotherapy and postoperative chemotherapy with fluorouracil and oxaliplatin versus fluorouracil alone in locally advanced rectal cancer: initial results of the German CAO/ARO/AIO-04 randomised phase 3 trial. Lancet Oncol. 2012 Jul;13(7):679-87. doi: 10.1016/S1470-2045(12)70187-0. Epub 2012 May 23. PMID 22627104
- [Background] Rodel F, Sprenger T, Kaina B, Liersch T, Rodel C, Fulda S, Hehlgans S. Survivin as a prognostic/predictive marker and molecular target in cancer therapy. Curr Med Chem. 2012;19(22):3679-88. doi: 10.2174/092986712801661040. PMID 22680927
- [Background] Sprenger T, Conradi LC, Beissbarth T, Ermert H, Homayounfar K, Middel P, Ruschoff J, Wolff HA, Schuler P, Ghadimi BM, Rodel C, Becker H, Rodel F, Liersch T. Enrichment of CD133-expressing cells in rectal cancers treated with preoperative radiochemotherapy is an independent marker for metastasis and survival. Cancer. 2013 Jan 1;119(1):26-35. doi: 10.1002/cncr.27703. Epub 2012 Jun 26. PMID 22736392
- [Background] Conradi LC, Styczen H, Sprenger T, Wolff HA, Rodel C, Nietert M, Homayounfar K, Gaedcke J, Kitz J, Talaulicar R, Becker H, Ghadimi M, Middel P, Beissbarth T, Ruschoff J, Liersch T. Frequency of HER-2 positivity in rectal cancer and prognosis. Am J Surg Pathol. 2013 Apr;37(4):522-31. doi: 10.1097/PAS.0b013e318272ff4d. PMID 23282976
- [Background] Wolff HA, Conradi LC, Beissbarth T, Leha A, Hohenberger W, Merkel S, Fietkau R, Raab HR, Tschmelitsch J, Hess CF, Becker H, Wittekind C, Sauer R, Rodel C, Liersch T; German Rectal Cancer Study Group. Gender affects acute organ toxicity during radiochemotherapy for rectal cancer: long-term results of the German CAO/ARO/AIO-94 phase III trial. Radiother Oncol. 2013 Jul;108(1):48-54. doi: 10.1016/j.radonc.2013.05.009. Epub 2013 Jun 11. PMID 23768685
- [Background] Sprenger T, Rothe H, Becker H, Beissbarth T, Homayounfar K, Gauss K, Kitz J, Wolff H, Scheel AH, Ghadimi M, Rodel C, Conradi LC, Liersch T. Lymph node metastases in rectal cancer after preoperative radiochemotherapy: impact of intramesorectal distribution and residual micrometastatic involvement. Am J Surg Pathol. 2013 Aug;37(8):1283-9. doi: 10.1097/PAS.0b013e3182886ced. PMID 23851331
- [Background] Fokas E, Conradi L, Weiss C, Sprenger T, Middel P, Rau T, Dellas K, Kitz J, Rodel F, Sauer R, Ruschoff J, Beissbarth T, Arnold D, Ghadimi BM, Rodel C, Liersch T. Preoperative chemoradiation therapy with capecitabine/oxaliplatin and cetuximab in rectal cancer: long-term results of a prospective phase 1/2 study. Int J Radiat Oncol Biol Phys. 2013 Dec 1;87(5):992-9. doi: 10.1016/j.ijrobp.2013.09.011. Epub 2013 Oct 24. PMID 24210078
- [Background] Quack H, Erpenbeck L, Wolff HA, Sprenger T, Seitz CS, Schon MP, Neumann S, Stanek K, Ghadimi BM, Michels B, Middel P, Schaefer IM, Liersch T, Conradi LC. Oxaliplatin-Induced Leukocytoclastic Vasculitis under Adjuvant Chemotherapy for Colorectal Cancer: Two Cases of a Rare Adverse Event. Case Rep Oncol. 2013 Dec 11;6(3):609-15. doi: 10.1159/000357166. eCollection 2013 Sep. PMID 24474925
- [Background] Folprecht G, Gruenberger T, Bechstein W, Raab HR, Weitz J, Lordick F, Hartmann JT, Stoehlmacher-Williams J, Lang H, Trarbach T, Liersch T, Ockert D, Jaeger D, Steger U, Suedhoff T, Rentsch A, Kohne CH. Survival of patients with initially unresectable colorectal liver metastases treated with FOLFOX/cetuximab or FOLFIRI/cetuximab in a multidisciplinary concept (CELIM study). Ann Oncol. 2014 May;25(5):1018-25. doi: 10.1093/annonc/mdu088. Epub 2014 Feb 27. PMID 24585720
- [Background] Fokas E, Liersch T, Fietkau R, Hohenberger W, Beissbarth T, Hess C, Becker H, Ghadimi M, Mrak K, Merkel S, Raab HR, Sauer R, Wittekind C, Rodel C. Tumor regression grading after preoperative chemoradiotherapy for locally advanced rectal carcinoma revisited: updated results of the CAO/ARO/AIO-94 trial. J Clin Oncol. 2014 May 20;32(15):1554-62. doi: 10.1200/JCO.2013.54.3769. Epub 2014 Apr 21. PMID 24752056
- [Background] Homayounfar K, Bleckmann A, Helms HJ, Lordick F, Ruschoff J, Conradi LC, Sprenger T, Ghadimi M, Liersch T. Discrepancies between medical oncologists and surgeons in assessment of resectability and indication for chemotherapy in patients with colorectal liver metastases. Br J Surg. 2014 Apr;101(5):550-7. doi: 10.1002/bjs.9436. Epub 2014 Feb 20. PMID 24756914
- [Background] Ilgen P, Stoldt S, Conradi LC, Wurm CA, Ruschoff J, Ghadimi BM, Liersch T, Jakobs S. STED super-resolution microscopy of clinical paraffin-embedded human rectal cancer tissue. PLoS One. 2014 Jul 15;9(7):e101563. doi: 10.1371/journal.pone.0101563. eCollection 2014. PMID 25025184
- [Background] Fokas E, Liersch T, Fietkau R, Hohenberger W, Hess C, Becker H, Sauer R, Wittekind C, Rodel C. Downstage migration after neoadjuvant chemoradiotherapy for rectal cancer: the reverse of the Will Rogers phenomenon? Cancer. 2015 Jun 1;121(11):1724-7. doi: 10.1002/cncr.29260. Epub 2015 Jan 21. PMID 25611452
- [Background] Scheel AH, Reineke RA, Sprenger T, Lokka S, Kitz J, Ghadimi BM, Ruschoff J, Liersch T, Middel P. Comprehensive lymph node morphometry in rectal cancer using acetone compression. J Clin Pathol. 2015 Jun;68(6):458-64. doi: 10.1136/jclinpath-2014-202555. Epub 2015 Mar 16. PMID 25779094
- [Background] Styczen H, Nagelmeier I, Beissbarth T, Nietert M, Homayounfar K, Sprenger T, Boczek U, Stanek K, Kitz J, Wolff HA, Ghadimi BM, Middel P, Liersch T, Ruschoff J, Conradi LC. HER-2 and HER-3 expression in liver metastases of patients with colorectal cancer. Oncotarget. 2015 Jun 20;6(17):15065-76. doi: 10.18632/oncotarget.3527. PMID 25915155
- [Background] Poschau M, Dickreuter E, Singh-Muller J, Zscheppang K, Eke I, Liersch T, Cordes N. EGFR and beta1-integrin targeting differentially affect colorectal carcinoma cell radiosensitivity and invasion. Radiother Oncol. 2015 Sep;116(3):510-6. doi: 10.1016/j.radonc.2015.06.005. Epub 2015 Jun 18. PMID 26096850
- [Background] Rodel C, Graeven U, Fietkau R, Hohenberger W, Hothorn T, Arnold D, Hofheinz RD, Ghadimi M, Wolff HA, Lang-Welzenbach M, Raab HR, Wittekind C, Strobel P, Staib L, Wilhelm M, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R, Liersch T; German Rectal Cancer Study Group. Oxaliplatin added to fluorouracil-based preoperative chemoradiotherapy and postoperative chemotherapy of locally advanced rectal cancer (the German CAO/ARO/AIO-04 study): final results of the multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2015 Aug;16(8):979-89. doi: 10.1016/S1470-2045(15)00159-X. Epub 2015 Jul 15. PMID 26189067
- [Background] Bleckmann A, Conradi LC, Menck K, Schmick NA, Schubert A, Rietkotter E, Arackal J, Middel P, Schambony A, Liersch T, Homayounfar K, Beissbarth T, Klemm F, Binder C, Pukrop T. beta-catenin-independent WNT signaling and Ki67 in contrast to the estrogen receptor status are prognostic and associated with poor prognosis in breast cancer liver metastases. Clin Exp Metastasis. 2016 Apr;33(4):309-23. doi: 10.1007/s10585-016-9780-3. Epub 2016 Feb 9. PMID 26862065
- [Background] Sprenger T, Rothe H, Conradi LC, Beissbarth T, Kauffels A, Kitz J, Homayounfar K, Wolff H, Strobel P, Ghadimi M, Wittekind C, Sauer R, Rodel C, Liersch T. Stage-Dependent Frequency of Lymph Node Metastases in Patients With Rectal Carcinoma After Preoperative Chemoradiation: Results from the CAO/ARO/AIO-94 Trial and From a Comparative Prospective Evaluation With Extensive Pathological Workup. Dis Colon Rectum. 2016 May;59(5):377-85. doi: 10.1097/DCR.0000000000000570. PMID 27050599
- [Background] Jo P, Nietert M, Gusky L, Kitz J, Conradi LC, Muller-Dornieden A, Schuler P, Wolff HA, Ruschoff J, Strobel P, Grade M, Liersch T, Beissbarth T, Ghadimi MB, Sax U, Gaedcke J. Neoadjuvant Therapy in Rectal Cancer - Biobanking of Preoperative Tumor Biopsies. Sci Rep. 2016 Oct 18;6:35589. doi: 10.1038/srep35589. PMID 27752113
- [Background] Sahlmann CO, Homayounfar K, Niessner M, Dyczkowski J, Conradi LC, Braulke F, Meller B, Beissbarth T, Ghadimi BM, Meller J, Goldenberg DM, Liersch T. Repeated adjuvant anti-CEA radioimmunotherapy after resection of colorectal liver metastases: Safety, feasibility, and long-term efficacy results of a prospective phase 2 study. Cancer. 2017 Feb 15;123(4):638-649. doi: 10.1002/cncr.30390. Epub 2016 Oct 20. PMID 27763687